CLINICAL TRIAL: NCT03998436
Title: A Prospective, Multicenter, Randomized, Double-Blind, Phase 3 Study to Evaluate the Safety and Efficacy of a Gel Formulation of Esmolol Hydrochloride (Galnobax®) in Treating Diabetic Foot Ulcers
Brief Title: Phase 3 Study to Evaluate the Safety and Efficacy of Galnobax® in Treating Diabetic Foot Ulcers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novalead Pharma Private Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NG-A16
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Results first posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-08

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — esmolol

STUDY DESIGN:
Intervention Model Description: Prospective, Multicenter, Randomized, Double-Blind, Parallel groups
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The subject will be masked from the treatment by the Study Nurse (care giver) by using blinder during each treatment application. The site has two separate teams (blinded and unblinded) for masking. The unblinded investigator performs application of treatment during each treatment visit of subject to the site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Galnobax® 14% gel plus SoC (Active Comparator): Galnobax 14% gel along with Standard of Care (SoC) will be administered twice daily (150 subjects)
  Interventions: Drug: Esmolol Hydrochloride
- SoC Only (Sham Comparator): Only Standard of Care will be administered twice daily (150 subjects)
  Interventions: Other: Only Standard of Care
- Vehicle plus SoC (Placebo Comparator): Vehicle gel along with Standard of Care (SoC) will be administered twice daily (50 subjects)
  Interventions: Other: Vehicle Gel

INTERVENTIONS:
Drug: Esmolol Hydrochloride — Galnobax-14% gel application along with Standard of Care
  Other Names: Galnobax
  Arms: Galnobax® 14% gel plus SoC
Other: Only Standard of Care — Only Standard of Care treatment
  Arms: SoC Only
Other: Vehicle Gel — Vehicle gel application along with Standard of Care
  Arms: Vehicle plus SoC

SUMMARY:
The purpose of the current Study is to determine the safety and effectiveness of Galnobax® plus Standard of Care versus only Standard of Care, in treating Diabetic Foot Ulcers (DFU). In addition, Study is designed to investigate the safety of Galnobax® vehicle for establishing non-deleterious effects of Vehicle on wound healing in the Subjects with DFU. The study is being conducted in 350 subjects being recruited in about 30 centers in India.

DETAILED DESCRIPTION:
The current study is a Prospective, Multicenter, Randomized, Double-Blind, Phase 3 Study to Evaluate the Safety and Efficacy of a Gel Formulation of Esmolol Hydrochloride (Galnobax®) in Treating Diabetic Foot Ulcers. The study evaluates the safety and effectiveness of Galnobax® plus Standard of Care versus only Standard of Care, in treating Diabetic Foot Ulcers (DFU). In addition, Study is designed to investigate the safety of Galnobax® vehicle for establishing non-deleterious effects of Vehicle on wound healing in the Subjects with DFU.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects, male or female, aged 18 to 75 years (inclusive) with Type 1 or Type 2 diabetes undergoing therapy for glycemic control
2. Subject has glycosylated hemoglobin, HbA1C, ≤ 12%
3. Subject with diagnosis of neuropathic foot ulcer by 10g monofilament test
4. Subject has adequate vascular perfusion of the affected limb, confirmed by Ankle-Brachial Index (ABI) ≥ 0.65 and ≤ 1.3
5. Presence of at least one DFU that meets all of the following criteria:

   1. A full-thickness ulcer of Grade A1 as per Texas classification system;
   2. Ulcer is located below or up to 5 cm above the malleoli (excluding ulcers between the toes);
   3. Ulcer size (area) is ≥ 2 cm2 and ≤ 15 cm2 (post-debridement);
   4. There is a minimum 3 cm margin between the qualifying Target Ulcer and any other ulcers on the specified foot, post-debridement;
   5. No exposed bone, tendon, muscle, ligament or joint capsule, and no tunneling, undermining, or sinus tracts;
   6. Unresponsive to ulcer care and open for at least 6 weeks at the time of the Screening Visit;
   7. Ulcer is non-infected as determined by clinical assessment and complete hemogram;
   8. Ulcer has a clean, granulating base free of adherent slough to the greatest extent possible as per Investigator;
   9. Ulcer area reduction < 30% from the Screening Visit to Baseline visit
6. Clinically normal resting 12-lead ECG at Screening Visit or, if abnormal, considered not clinically significant by the Investigator
7. Subject, if female of child-bearing potential, has a negative urine pregnancy test at Screening and willing to use acceptable methods of contraception (birth control pills, barriers) or abstinence throughout the Study
8. Subject is able and willing to comply with Study procedures including the use of an off-loading device (as applicable for the location of the ulcer) and adhere to protocol during the Study in the opinion of Investigator
9. A Subject or LAR agrees to sign informed consent form and allow audio visual recording of consent, if applicable

Exclusion Criteria:

1. Actively infected ulcers with or without purulent discharge, ulcers with exposed bone or associated with osteomyelitis
2. Subjects with more than three ulcers below knee
3. Subjects with Target Ulcer requiring off-loading that cannot be effectively off-loaded; or unable to tolerate the off-loading method
4. Subject has ulcers caused by a disease other than diabetes, e.g., fungal ulcerations, malignant ulcerations, and ulcerations due to venous or arterial insufficiency, or due to hematological disorders, in the opinion of the Investigator
5. Ulcer, about which the Investigator is suspicious for cancer
6. Subjects with a gangrenous or ischemic ulcer
7. Subject with ulcer that in the opinion of the Investigator, may need amputation
8. Subject with Target ulcer where wound measurement is not possible, such as ulcers between toes
9. Body mass index (BMI) > 40 kg/m2
10. Laboratory values at Screening of:

    1. Hemoglobin < 10.0 g/dL
    2. White Blood Cells (WBC) < 2.0 X 109 cells/L
    3. Liver function studies [Total bilirubin, aspartate aminotransferase (AST) and alanine transaminase (ALT)] > 3x the upper limit of normal
    4. Albumin < 2.5 g/dL
    5. eGFR < 25 mL/min
11. Presence of any existing clinically significant medical condition(s) that, in the opinion of the Investigator, could interfere with wound healing
12. Subject has received or is currently receiving or scheduled to receive any medication or therapies during the course of the Study that will modulate wound healing
13. Subject with intolerance to β-blockers at any time in the past
14. Has any other factor which may, in the opinion of the Investigator, compromise participation and/or follow-up in the Study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2018-12-26 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashu Rastogi, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (14):
- India (14):
  - Yalamanchi Hospita, Vijayawada, Andhra Pradesh
  - M.S. Ramaiah Medical College and Hospital, Bangalore, Karnataka
  - Sapthagiri Institute of Medical Sciences and Research Centre, Bangalore, Karnataka
  - Rajlaxmi Hospital, Bangalore, Karnataka
  - Sri Siddhartha Medical College, Tumkūr, Karnataka
  - Sujata Birla Hospital & Medical Research Center, Nashik, Maharashtra
  - Deenanath Mangeshkar Hospital and Research Center, Pune, Maharashtra
  - Chellaram Diabetes Institute, Pune, Maharashtra
  - Appollo Hospital, Chennai, Tamil Nadu
  - M.V. Hospital for Diabetes Pvt Ltd, Chennai, Tamil Nadu
  - Madras Diabetes Research Foundation, Chennai, Tamil Nadu
  - Sri Ramachandra Hospital, Chennai, Tamil Nadu
  - Post Graduate Institute of Medical Education and Research (PGIMER), Chandigarh
  - Maharaja Agrasen Hospital, New Delhi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rastogi A, Kulkarni SA, Agarwal S, Akhtar M, Arsule S, Bhamre S, Bhosle D, Desai S, Deshmukh M, Giriraja KV, Jagannath J, Kashiva RY, Kesavan R, Khandelwal D, Kolte S, Kongara S, Darivemula AK, Madhusudan C, Pyare Saheb Qureshi MAH, Ramu M, Rathod G, Yalamanchi SR, Shakya S, Shetty P, Singh S, Deshpande SK, Viswanathan V, Unnikrishnan AG. Topical Esmolol Hydrochloride as a Novel Treatment Modality for Diabetic Foot Ulcers: A Phase 3 Randomized Clinical Trial. JAMA Netw Open. 2023 May 1;6(5):e2311509. doi: 10.1001/jamanetworkopen.2023.11509. PMID 37184839

RESULTS

PARTICIPANT FLOW:
Groups:
- Galnobax® 14% Gel Plus SoC: Esmolol Hydrochloride gel (Galnobax) administered twice daily along with Standard of Care
- SoC Only: Only Standard of Care administered twice daily
- Vehicle Plus SoC: Vehicle gel administered twice daily along with Standard of Care
Period: Overall Study
Arm/Group | Galnobax® 14% Gel Plus SoC | SoC Only | Vehicle Plus SoC
Started | 76 | 76 | 24
Completed | 68 | 72 | 23
Not Completed | 8 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Galnobax® 14% Gel Plus SoC | SoC Only | Vehicle Plus SoC | Total
Number analyzed (Participants) | 76 | 76 | 24 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (8.96) | 56.1 (9.36) | 57.3 (8.01) | 56.4 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 9 | 54
  Male | 55 | 52 | 15 | 122
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  India | 76 | 76 | 24 | 176
Body Mass Index [Mean (Standard Deviation); unit: Kg/m2] | 26.7 (4.05) | 25.9 (4.30) | 25.9 (3.39) | 26.2 (4.08)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving Target Ulcer Closure Within 12-week Treatment Phase, as Assessed by Blinded Investigator
Description: Proportion of complete closure of wounds within 12-week treatment phase where Complete wound closure is defined as complete skin re-epithelialization that is without drainage or dressing requirements evaluated in two visits two weeks apart from first observation of closure.
Time Frame: Wound closure assessed up to week 12 and confirmed by 2 visits 2 weeks apart; only participants with wound closure at or before Week 12 and who maintained closure after 4-weeks of follow-up reported
Population: Subjects in FAS population
Measure: Count of Participants; unit: Participants
Arm/Group | Galnobax® 14% Gel Plus SoC | SoC Only | Vehicle Plus SoC
Number analyzed (Participants) | 68 | 72 | 23
Participants | 41 | 30 | 10
Statistical Analysis 1: Comparison: Galnobax® 14% Gel Plus SoC vs SoC Only; Test type: Superiority; p = 0.0276, Chi-squared; Odds Ratio (OR) = 2.126, 95% CI 2-sided [1.08 to 4.17]

2. Secondary Outcome: Proportion of Subjects Achieving Target Ulcer Closure Till End of Study, as Assessed by the Blinded Investigator.
Description: Proportion of complete closure of wounds at 24-weeks or End of Study where Complete wound closure is defined as complete skin re-epithelialization that is without drainage or dressing requirements.
Time Frame: 24-weeks. The ulcers achieving complete closure till end of study
Measure: Count of Participants; unit: Participants
Arm/Group | Galnobax® 14% Gel Plus SoC | SoC Only | Vehicle Plus SoC
Number analyzed (Participants) | 57 | 63 | 23
Participants | 44 | 35 | 9
Statistical Analysis 1: Comparison: Galnobax® 14% Gel Plus SoC vs SoC Only; Test type: Superiority; p = 0.0126, Chi-squared; Odds Ratio (OR) = 2.708, 95% CI 2-sided [1.22 to 5.99]

3. Other Pre Specified Outcome: Proportion of Subjects With Treatment Emergent Adverse Events (TEAEs)
Description: Proportion of Treatment emergent adverse events (TEAEs) in all the groups
Time Frame: 24-weeks
Population: ITT (Safety population)
Measure: Count of Participants; unit: Participants
Arm/Group | Galnobax® 14% Gel Plus SoC | SoC Only | Vehicle Plus SoC
Number analyzed (Participants) | 76 | 76 | 24
Participants | 10 | 14 | 9

ADVERSE EVENTS:
Time Frame: 24 weeks i.e. till end of study
Description: AEs collected from baseline visit i.e. after first application of treatment
Groups:
- Galnobax® 14% Gel Plus SoC: Galnobax 14% gel along with Standard of Care (SoC) will be administered twice daily (76 subjects)
  Esmolol Hydrochloride: Galnobax-14% gel application along with Standard of Care
- SoC Only: Only Standard of Care will be administered twice daily (76 subjects)
  Only Standard of Care: Only Standard of Care treatment
- Vehicle Plus SoC: Vehicle gel along with Standard of Care (SoC) will be administered twice daily (24 subjects)
  Vehicle Gel: Vehicle gel application along with Standard of Care
Arm/Group | Galnobax® 14% Gel Plus SoC | SoC Only | Vehicle Plus SoC
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/76 | 1/24
Serious Adverse Events (participants affected / at risk) | 1/76 | 2/76 | 4/24
Other Adverse Events (participants affected / at risk) | 9/76 | 7/76 | 9/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galnobax® 14% Gel Plus SoC (N=76) | SoC Only (N=76) | Vehicle Plus SoC (N=24)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galnobax® 14% Gel Plus SoC (N=76) | SoC Only (N=76) | Vehicle Plus SoC (N=24)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 5 (5) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

The sponsor has prepared an integrated clinical/statistical report. As this was a multicenter study, any publication/presentation of data was to include the entire study population. Publication/presentation of data from individual study centers is not allowed without explicit permission from the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-28): https://cdn.clinicaltrials.gov/large-docs/36/NCT03998436/Prot_SAP_000.pdf